CLINICAL TRIAL: NCT02610842
Title: Hands on - a Hand Care Guide in Systemic Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Eduardo de Paiva Magalhães, MD, PhD, University of Campinas, Brazil
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UOP01
Record Dates: First submitted 2015-11-12; First posted 2015-11-20 (Estimated); Results first posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-01

CONDITIONS: Scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Handbook group (Experimental): Patients will receive a home based program named "Hands on" - a hand care guide in Systemic Sclerosis" which includes a handbook with instructions about the disease and hand exercises. Patients will be asked to follow the program instructions and carry out the exercises daily during the following 12 weeks.
  Interventions: Other: Handbook

INTERVENTIONS:
Other: Handbook — The handbook named "Hands on" - a hand care guide in Systemic Sclerosis" contains instructions about the Systemic Sclerosis and hand exercises.

SUMMARY:
Hands are commonly affected in Systemic Sclerosis (SS). The objective of this research is to apply a home based hand care guide in patients with SS and to evaluate its response regarding hand pain, function, strength and mobility.

DETAILED DESCRIPTION:
Introduction: Hands are commonly affected in Systemic sclerosis (SS). Skin thickening, Raynaud phenomenon, digital ulcers and cutaneous calcinosis may result in pain, disability and claw deformity. Strategies to improve hand function are recommended since its diagnosis and throughout the treatment. Unfortunately hand care assistance is not often available. The objective of this study was to developed a brief guide about hand care and home-based exercises to be applied in our outpatient clinic.

Methods: A brief program , with instructions about the disease and home-based exercises will be applied in a group patients with Systemic Sclerosis (SS) during the period of 12 weeks. Hand function (Cochin Hand and Functional Scale), disability (HAQ-Scleroderma), quality of life (SF-36 hand pain (visual analogue scale), grip and pinch strength, hand mobility (delta finger) will be assessed in the first appointment and after twelve weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Systemic Scleroderma according to the American College of Rheumatology (Criteria Committee, Arthritis Rheum. 2013).
* Involvement of hands with skin thickening.
* Interest in participating in the investigation
* Ability to read and to answer the the proposed questionnaires

Exclusion Criteria:

* Upper limb commitment due other reasons other than Systemic Sclerosis.
* Presence of digital ulcers, hand deformities or conditins that impede the realization of the proposed exercises
* Clinical manifestations that impede the performance of the proposed exercises

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bertolo B Manoel, MD,PhD, Study Director — University of Campinas
Locations (2):
- Brazil (2):
  - Clinical Hospital of University of Campinas, Campinas, São Paulo
  - University of Campinas, Campinas, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Subjects baseline characteristics are shown in results (age,

REFERENCES:
- [Background] Mayes MD. Scleroderma epidemiology. Rheum Dis Clin North Am. 2003 May;29(2):239-54. doi: 10.1016/s0889-857x(03)00022-x. PMID 12841293
- [Background] Skare TL, Toebe BL, Boros C. Hand dysfunction in scleroderma patients. Sao Paulo Med J. 2011;129(5):357-60. doi: 10.1590/s1516-31802011000500012. No abstract available. PMID 22069136
- [Background] Torok KS, Baker NA, Lucas M, Domsic RT, Boudreau R, Medsger TA Jr. Reliability and validity of the delta finger-to-palm (FTP), a new measure of finger range of motion in systemic sclerosis. Clin Exp Rheumatol. 2010 Mar-Apr;28(2 Suppl 58):S28-36. Epub 2010 Jun 10. PMID 20576211

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with SSc were invited to take part in this study during their routine appointments at University of Campinas Rheumatology Outpatient Clinic.
Pre-assignment Details: Patients were excluded if enrolled in other rehabilitation program in the previous three months, in the presence of hand disability due other pathologies rather than Systemic Sclerosis, or if they could not perform the exercises proposed as intevention due to medical conditions or advanced hand deformities.
Period: Overall Study
Arm/Group | Handbook Group
Started | 27
Completed | 22
Not Completed | 5
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Groups:
- Handbook Group: Patients with systemic scleroderma and hands commitment.
Arm/Group | Handbook Group
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 5 subjects did not complete the protocol and were not used for analysis
  years
    number analyzed (Participants) | 22
    (all) | 48.09 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 5 subjects did not complete the protocol and were not used for analysis
  Participants
    number analyzed (Participants) | 22
    Female | 18
    Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 5 subjects did not complete the protocol and were not used for analysis
  Participants
    number analyzed (Participants) | 22
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 13
    More than one race | 9
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 22

OUTCOME MEASURES:

1. Primary Outcome: Cochin Hand Functional Scale
Description: The purpose of this self-report scale is to measure functional ability in the hand.
  The questions ask how much difficulty the person has performing 18 tasks without the help of any assistive device. Kitchen tasks include holding a bowl and a plate full of food, pouring liquid, cutting meat, and peeling fruit. The dressing items include buttoning and opening/closing a zipper. The hygiene items include squeezing a tube of toothpaste and holding a toothbrush. Office items include 2 writing tasks, while other items include turning a doorknob, cutting with scissors, and turning a key in a lock. Score range is from 0-90. A higher score indicates greater disability or more difficulty, whereas a lower score indicates less disability or difficulty.
Time Frame: 08 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Handbook Group: Systemic Scleroderma subjects
Arm/Group | Handbook Group
Number analyzed (Participants) | 22
units on a scale | 19.24 (15.78)

2. Primary Outcome: Visual Analogue Pain Scale
Description: Hand pain (pain-VAS) was assessed using a 10 cm horizontal pain scale. Pain severity was rated from 0-10, where 0 = no pain and 10 = very severe pain
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Handbook Group: Systemic Sclerosis subjects
Arm/Group | Handbook Group
Number analyzed (Participants) | 22
units on a scale | 3.97 (4.5)

3. Secondary Outcome: Delta Finger-to-palm
Description: The standard finger-to-palm (FTP) measurement is obtained using a ruler to measure the distance (in centimeters)between the tip of the pulp on the 3rd finger and the distal palmar crease while the patient attempts to make a full fist (maximal finger flexion at all 3 finger joints: MCP, PIP, and DIP). The delta FTP is finger extension, the distance between the 3rd fingertip and the distal palmar crease while the patient attempts full finger extension, minus the FTP.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Handbook Group
Number analyzed (Participants) | 22
Centimeters | 92.86 (34.7)

4. Secondary Outcome: Scleroderma Health Assessment Questionnaire
Description: The Health Assessment Questionnaire, is a self-administered 20-questionnaire that assesses functional ability in eight domains. Questions in each domain are scored in a four-point scale, from 0 ("without difficulty") to 3 ("unable to do"). The maximum score from each domain is added together and divided by the number of categories completed (score ranging from 0 -better to 3 - worse). The Scleroderma Health Assessment Questionnaire (SHAQ) consists of the 20 items from the HAQ and has five additional questions that assess symptoms caused by Systemic Sclerosis (Raynaud Phemonomenon, digital tip ulcers, gastrointestinal and lung symptoms, as well as overall disease symptoms) using visual analogue scales (VAS). Scores on the VAS range from 0 (does not interfere with activities) to 3 (very severe limitations with activities). The overall score is the sum of each of the five VAS sub scores and the scores for the eight HAQ domains divided by 13. The SHAQ index ranges from 0 to 3.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Handbook Group
Number analyzed (Participants) | 22
units on a scale | 0.95 (0.53)

ADVERSE EVENTS:
Arm/Group | Handbook Group
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less